CLINICAL TRIAL: NCT06791226
Title: Evaluating the Potential Usefulness of 18F-AlF-FAPI PET/ CT in Patients With Orbital Neoplasms and Compared With 18F-FDG PET/ CT
Brief Title: Evaluating the Usefulness of 18F-AlF-FAPI PET/ CT in Orbital Neoplasms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: FAPI-Orbital Neoplasms
Record Dates: First submitted 2024-04-07; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Orbital Neoplasms
MeSH Terms: conditions — Orbital Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental): Experimental arm
  Interventions: Diagnostic Test: 18F-AlF-FAPI PET/CT, 18F-FDG PET/CT

INTERVENTIONS:
Diagnostic Test: 18F-AlF-FAPI PET/CT, 18F-FDG PET/CT — Subjects with orbital neoplasms underwent contemporaneous 18F-AlF-FAPI and 18F-FDG PET/CT for diagnosis and staging.

SUMMARY:
To evaluate the potential usefulness of 18F-AlF-FAPI positron emission tomography/computed tomography (PET/CT) for the diagnosis of primary and metastatic lesions in orbital neoplasms, and compared with 18F-FDG PET/CT.

DETAILED DESCRIPTION:
Subjects with orbital neoplasms underwent contemporaneous 18F-AlF-FAPI and 18F-FDG PET/CT for initial assessment. Tumor uptake was quantified by the maximum standard uptake value (SUVmax). The numbers of metastatic lesions of 18F-FDG and 18F-AlF-FAPI PET/CT were recorded by visual interpretation. The sensitivity, specificity, and accuracy of 18F-AlF-FAPI, 18F-FDG PET/CT were calculated and compared to evaluate the diagnostic accuracy.

ELIGIBILITY:
Inclusion Criteria:

1. patients with suspected or newly diagnosed orbital neoplasms (supporting evidence may include MRI, CT and pathology report);
2. patients who had scheduled both 18F-FDG and 18F-AlF-FAPI PET/CT scans;
3. patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

1. patients with pregnancy;
2. breastfeeding;
3. the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 3 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-07-16 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy | through study completion, an average of 6 months
  The diagnostic accuracy of 18F-FDG and 18F-AlF-FAPI PET/CT were calculated and compared to evaluate the diagnostic efficacy.

SECONDARY OUTCOMES:
SUV metrics | through study completion, an average of 6 months
  Standardized uptake value (SUV) metrics of 18F-FDG and 18F-AlF-FAPI PET/CT for each target lesion of subject or suspected primary tumor or/and metastasis.
Tumor-to-background ratio | through study completion, an average of 6 months
  tumor-to-background ratio of 18F-FDG and 18F-AlF-FAPI PET/CT for each target lesion of subject or suspected primary tumor or/and metastasis.
Number of lesions | through study completion, an average of 6 months
  The numbers of positive primary and metastatic lesions of 18F-FDG and 18F-AlF-FAPI PET/CT were recorded by visual interpretation.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Nuclear Medicine, Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No